CLINICAL TRIAL: NCT02597517
Title: Optical Enhancement System ™ Plus Optical Magnification Utility in the Identification of Normal Gastric Mucosa, Helicobacter Pylori Associated Gastritis, and Gastric Atrophy
Brief Title: New Technology to Differentiate Normal Gastric Mucosa From Helicobacter Pylori Associated Gastritis and Gastric Atrophy
Status: Completed | Type: Observational
Sponsor: Instituto Ecuatoriano de Enfermedades Digestivas (Other)
Responsible Party: Sponsor
Other Study IDs: Sept-1-2015
Record Dates: First submitted 2015-10-19; First posted 2015-11-05 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-05

CONDITIONS: Gastritis; Helicobacter Pylori Associated Gastritis; Atrophic Gastritis
Keywords: gastritis; chromoendoscopy; magnification; Helicobacter pylori; Atrophic gastritis
MeSH Terms: conditions — Gastritis; Gastritis, Atrophic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Histological biopsies from gastric mucosal
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Intervention group: (Digital chromoendoscopy and magnification) Patients with functional dyspepsia and positive stool antigen test for H pylori in whom gastric body mucosal will be evaluated with digital chromoendoscopy (OE system) and magnification technology in addition to white light
  Interventions: Device: Digital chromoendoscopy and magnification
- Control group: (Digital chromoendoscopy and magnification) Patients with functional dyspepsia and negative stool antigen test for H pylori in whom gastric mucosal body will be evaluated with digital chromoendoscopy (OE system) and magnification technology in addition to white light
  Interventions: Device: Digital chromoendoscopy and magnification

INTERVENTIONS:
Device: Digital chromoendoscopy and magnification — After the gastric body mucosal evaluation with white light endoscopy, the Optical Enhancement chromoendoscopy and magnification will be used for a more detailed evaluation of the subepithelial capillary network, the collecting venules and mucosal pits
  Other Names: OE System (EPK-i7010) and Magniview (EG-2990Zi)

SUMMARY:
Endoscopy is a tool that has greatly influenced gastroenterological diagnosis. However, conventional endoscopy is limited to detecting lesions on the basis of gross morphological changes and therefore a certainly diagnosis depends on biopsy sampling of macroscopically obvious endoscopic features, or blind biopsy sampling of normal appearing mucosa with the risk of missed pathology and sampling errors.

Gastric cancer is the second most common cause of cancer related death. One of the main roles of upper gastrointestinal endoscopy is to identify gastric cancer at an early stage. The importance of identifying H. pylori infection is because it plays a very important role in gastric carcinogenesis, progressing from chronic gastritis through atrophic gastritis, intestinal metaplasia, dysplasia and finally cancer. The importance of recognition a precancerous gastric lesion is because we can detect most tumors at an early stage and improve the survival.

Most studies conclude that it is difficult to diagnose H. pylori related gastritis and gastric atrophy on the basis of endoscopic findings. Histology is therefore currently considered to be the gold standard for detecting H. pylori infection. The reliability of detecting H. pylori infection histologically depends on the site, number, and size of gastric biopsy specimens, as well as on expertise in staining and visualizing the bacteria. Considerable error also occurs in identifying gastric atrophy using blind biopsy sampling, and neither the original nor the revised version of the Sydney system reliably identifies more than half the cases in patients with confirmed gastric atrophy.

DETAILED DESCRIPTION:
Recently an image-enhanced endoscopic technology using a pre-processor band-limited light called Optical Enhancement system (OE system™), was developed by HOYA Co. (Tokyo, Japan) and is now equipped with the latest endoscopy system (Pentax Video Processor EPK-i7010; HOYA Co.). This new technology combines digital signal processing in a similar way to I-scan and optical filters that limit the spectral characteristics of the illumination light. Previous I-scan technology uses white light alone as an illumination light and digital post-processing of the reflection afterwards creates images yielding the virtual chromoendoscopic image. Emission of white light alone causes a potential limitation for the current I-scan technology to obtain higher contrast images of microvascular pattern on the mucosal surface in combination with high magnification as shown by NBI with optical magnification. The basic concept of OE is to overcome the darkness of NBI witch results in less usefulness for detectability in wide-range observation in the gastrointestinal lumen. The new innovated optical filters achieve higher overall transmittance by connecting the peaks of the hemoglobin absorption spectrum (415 nm, 540 nm and 570 nm) creating a continuous wavelength spectrum. There are two modes with different OE filters (Mode 1 and Mode 2). Mode 1 is designed mainly to improve visualization of microvessels with a sufficient amount of light, and Mode 2 is designed to improve contrast of white-light observation by bringing the color tone of the overall image closer to that of natural color (white color tone) with much more light than that of the Mode 1 filter.

In addition to this, new scopes have been developed which combines high definition images with optical magnification called Magniview™. These scopes increase the image up to 136 times with a better quality of image than standard scopes without optical zoom. This allows an optimal and much clear evaluation of the mucosa and superficial vascular aspects, possibly identifying early suggestive signs of inflammation or lesions not seen before using conventional videoendoscopy, high definition scopes with white light or digital post-processor filters systems as I-Scan™.

Estimated enrollment: A total of 100 patients with functional dyspepsia will be include (intervention group: 50 patients and control group: 50 patients)

Study design: This is an observational and analytical cross-section, population - based survey study, with a prospective case collection, non randomized and double blind, performed in a Tertiary Academic Center.

* Allocation: Non randomized, double blind
* Endpoint Classification: Efficacy
* Intervention Model: Non interventional
* Primary Purpose: Diagnosis

Setting: Ecuadorian Institute of Digestive Diseases (IECED), OmniHospital Academic Tertiary Center. We will include patients from October 2015 to December 2015. Patients will be recruited from the gastroenterology unit (IECED). The study protocol and consent form has been approved by the Institutional Review Board (IRB) and will be conducted according to the declaration of Helsinki. Patients will sign an informed consent.

Population selection, inclusion and exclusion criteria: All of the participants with functional dyspepsia will be tested for Helicobacter Pylori (HP) using the stool antigen test. After this phase we will have to groups of patients, dyspeptic HP (+) and dyspeptic HP (-). The first group will be the intervention group and the dyspeptic HP (-) patients will serve as control group. None the patients or the endoscopist will know which group each patient belongs.

Functional dyspepsia will be considered according to the Rome III. Criteria. It will include Epigastric pain Syndrome defined as located pain or burning in the upper abdomen, at least once a week, intermittent, not generalized, not relieved by defecation and without criteria of gall bladder or sphincter of Oddi pathology; and Postprandial distress Syndrome defined as the presence of one or both conditions including nagging feeling of postprandial fullness after normal volume meals, several times a week and early satiety that prevents the completion of a regular meal, several times a week. The criteria must be present in the last three months and have started at least 6 months before diagnosis.

Endoscopic technique: All the patients included in the protocol (intervention group and control group) will be studied by upper endoscopy with Magniview™ scopes and EPK-i7010 processor (OE system™). The endoscopy images will be seen on a 27inch, flat panel, high definition LCD monitor (Radiance™ ultra SC-WU27-G1520 model). The endoscopies will be performed by three endoscopist trained on this new technology (all of them with more than 10 procedures).

Initially a complete (esophagus, stomach, duodenum) conventional white light upper endoscopy will be performed with detailed observation of the whole stomach. After this the gastric body will be evaluated with the OE System and Magniview.

The technique involves the use of a distal black rubber hood (OE-A58) at the tip of the scope (EG-2990Zi) to fix the distance between the tip of the endoscope and the gastric mucosa at 2mm. First the OE system™ will be used (mode 1 and 2), then the optical magnification will be implemented through the actions of a button on the Magniview scope. After reaching the maximum magnification level, the cup will contact to the gastric mucosa and water will be instilled.

Any residue in the stomach will be removed using a water ejection pump. The evaluation of the gastric mucosa will be performed in the gastric body instead of the antrum because in the antrum the collecting venules lie in deeper layers and cannot be seen.

The endoscopic findings in the gastric body will be classified as the Anagnostopoulos GK et al. classification into four types: type 1, honeycomb-type subepithelial capillary network (SECN) with regular arrangement of collecting venules and regular, round pits; type 2, honeycomb-type SECN with regular, round pits, but loss of collecting venules; type 3, loss of normal SECN and collecting venules, with enlarged white pits surrounded by erythema; and type 4, loss of normal SECN and round pits, with irregular arrangement of collecting venules. Type 1 pattern for predicting normal gastric, types 2 and 3 patterns for predicting a Helicobacter pylori infection and type 4 patterns for predicting gastric atrophy.

The gastric body will be photographically recorded, including images of normal mucosa or gastric mucosal changes. Finally biopsies will be taken in both groups, using a regular biopsy forceps; randomly biopsies following the Sydney protocol (two from the gastric body, two from the antrum and one from the incisura angularis) and targeted biopsies from areas with a type 2,3 or 4 pattern, to correlate them with the histological changes in H. pylori gastritis and gastric atrophy. The diagnosis of positive H. pylori infection will be done to all participants by direct visualization at histological examination and using a stool antigen test for H pylori.

Interobserver and Intraobserver Agreement: A data set containing photographs of the gastric lesions will be presented to three blinded endoscopists who will confirm or not the findings. Inter and intra-observer reproducibility will be measured based on comparison of still images between the three investigators. To evaluate the intra-observer agreement each investigator will assess the images two times and the answers will be compared. To evaluate the inter-observer agreement all answers between the three investigators will be compared.

Statistical analysis: Base line characteristics will be compared between case and control group using Chi-square o Fisher Test for categorical variable, and for continuing variables, the Mann-Whitney Test will be used. The sensitivity, specificity, and predictive values of the endoscopic findings for normal gastric mucosa, H. pylori infection, and gastric atrophy will be calculated. To examine inter and intra observer agreement, kappa values will be calculated. A P value of less than 0.05 is considered to be statistically significant. All the statistical analysis will be performed using SPSS software suite v.22.

Limitations: The protocol will be performed in only one center and the group selection is not random

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years old patients
* Who agree to participate in the study
* Patients with functional dyspeptic symptoms

Exclusion Criteria:

* Patients, who were receiving nonsteroidal anti-inflammatory drugs, pump inhibitors (PPI) or antibiotics in the last 3 weeks.
* Severe uncontrolled coagulopathy
* Prior history of gastric surgery.
* Pregnancy and lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Two groups of functional dyspeptic patients will be selected randomly. Functional dyspepsia will be considered according to the Rome III. Criteria. It will include Epigastric pain Syndrome defined as located pain or burning in the upper abdomen, at least once a week, intermittent, not generalized, not relieved by defecation and without criteria of gall bladder or sphincter of Oddi pathology; and Postprandial distress Syndrome defined as the presence of one or both conditions including nagging feeling of postprandial fullness after normal volume meals, several times a week and early satiety that prevents the completion of a regular meal, several times a week. The criteria must be present in the last three months and have started at least 6 months before diagnosis.
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2015-11; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Utility OE System™ + Magniview™ in the diagnosis of normal gastric mucosa. Number of patients with type 1 in the Anagnostopoulos GK et al. classification. | two months
  Anagnostopoulos GK et al. classified the gastric body mucosal in four types: type 1, honeycomb-type subepithelial capillary network (SECN) with regular arrangement of collecting venules and regular, round pits. Type 1 pattern for predicting normal gastric mucosa.
Utility OE System™ + Magniview™ in the diagnosis of Helicobacter pylori associated gastritis. Number of patients with type 2,3 in the Anagnostopoulos GK et al. classification. | two months
  Anagnostopoulos GK et al. classified the gastric body mucosal in four types: type 2, honeycomb-type SECN with regular, round pits, but loss of collecting venules; type 3, loss of normal SECN and collecting venules, with enlarged white pits surrounded by erythema. Types 2 and 3 patterns for predicting a Helicobacter pylori infection.
Utility OE System™ + Magniview™ in the diagnosis of gastric atrophy. Number of patients with type 4 in the Anagnostopoulos GK et al. classification. | two months
  Anagnostopoulos GK et al. classified the gastric body mucosal in four types: type 4, loss of normal SECN and round pits, with irregular arrangement of collecting venules. Type 4 patterns for predicting gastric atrophy.

SECONDARY OUTCOMES:
Measures inter and intra-observer reproducibility in the assessment of the endoscopic patterns detected. | two months
  A data set containing photographs of the gastric lesions will be presented to three blinded endoscopists who will confirm or not the findings. Inter and intra-observer reproducibility will be measured based on comparison of still images between the three investigators. To evaluate the intra-observer agreement each investigator will assess the images three times and the answers will be compared. To evaluate the inter-observer agreement all answers between the three investigators will be compared. To examine inter and intra observer agreement, kappa values will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Robles-Medranda, MD, Principal Investigator — Ecuadorian Institute of Digestive Diseases
Locations (1):
- Instituto Ecuatoriano de Enfermedades Digestivas, Omnihospital, Guayaquil, Guayas, Ecuador

REFERENCES:
- [Result] Anagnostopoulos GK, Yao K, Kaye P, Fogden E, Fortun P, Shonde A, Foley S, Sunil S, Atherton JJ, Hawkey C, Ragunath K. High-resolution magnification endoscopy can reliably identify normal gastric mucosa, Helicobacter pylori-associated gastritis, and gastric atrophy. Endoscopy. 2007 Mar;39(3):202-7. doi: 10.1055/s-2006-945056. Epub 2007 Feb 1. PMID 17273960
- [Result] Correa P. Human gastric carcinogenesis: a multistep and multifactorial process--First American Cancer Society Award Lecture on Cancer Epidemiology and Prevention. Cancer Res. 1992 Dec 15;52(24):6735-40. PMID 1458460
- [Result] Whiting JL, Sigurdsson A, Rowlands DC, Hallissey MT, Fielding JW. The long term results of endoscopic surveillance of premalignant gastric lesions. Gut. 2002 Mar;50(3):378-81. doi: 10.1136/gut.50.3.378. PMID 11839718
- [Result] Bah A, Saraga E, Armstrong D, Vouillamoz D, Dorta G, Duroux P, Weber B, Froehlich F, Blum AL, Schnegg JF. Endoscopic features of Helicobacter pylori-related gastritis. Endoscopy. 1995 Oct;27(8):593-6. doi: 10.1055/s-2007-1005764. PMID 8608753
- [Result] Calabrese C, Di Febo G, Brandi G, Morselli-Labate AM, Areni A, Scialpi C, Biasco G, Miglioli M. Correlation between endoscopic features of gastric antrum, histology and Helicobacter pylori infection in adults. Ital J Gastroenterol Hepatol. 1999 Jun-Jul;31(5):359-65. PMID 10470592
- [Result] Dixon MF, Genta RM, Yardley JH, Correa P. Classification and grading of gastritis. The updated Sydney System. International Workshop on the Histopathology of Gastritis, Houston 1994. Am J Surg Pathol. 1996 Oct;20(10):1161-81. doi: 10.1097/00000478-199610000-00001. PMID 8827022
- [Result] Neumann H, Fujishiro M, Wilcox CM, Monkemuller K. Present and future perspectives of virtual chromoendoscopy with i-scan and optical enhancement technology. Dig Endosc. 2014 Jan;26 Suppl 1:43-51. doi: 10.1111/den.12190. Epub 2013 Oct 23. PMID 24373000
- [Result] Drossman DA. The functional gastrointestinal disorders and the Rome III process. Gastroenterology. 2006 Apr;130(5):1377-90. doi: 10.1053/j.gastro.2006.03.008. No abstract available. PMID 16678553